CLINICAL TRIAL: NCT03817502
Title: A 6-week, International, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of the Efficacy and Safety of Cariprazine in the Treatment of Adolescent Participants (13 to 17 Years of Age) With Schizophrenia
Brief Title: Efficacy and Safety of Cariprazine in the Treatment of Adolescent Participants (13 to 17 Years of Age) With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RGH-MD-20; 2018-004006-26 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cariprazine 1.5 mg/d (Experimental): Cariprazine capsules, oral administration, once daily.
  Interventions: Drug: Cariprazine
- Cariprazine 4.5 mg/d (Experimental): Cariprazine capsules, oral administration, once daily.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Matching placebo capsules, oral administration, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Cariprazine capsules, oral administration, once daily.
  Arms: Cariprazine 1.5 mg/d; Cariprazine 4.5 mg/d
Drug: Placebo — Matching placebo capsules, oral administration, once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cariprazine in the treatment of schizophrenia in the adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 primary diagnosis of schizophrenia.
* Schizophrenia diagnosis confirmed by the K-SADS-PL administered at screening (Visit 1) by a trained clinician.
* PANSS score ≥ 70 and a score of ≥ 4 (moderate) on 2 or more of the 5 items on the positive subscale of the PANSS (delusions, conceptual disorganization, hallucinatory behavior, grandiosity, suspiciousness/persecution), at screening (Visit 1) and baseline (Visit 2).
* CGI-S scale score of ≥ 4 (moderately ill) at screening (Visit 1) and baseline (Visit 2).

Exclusion Criteria:

* Current diagnosis of bipolar disorder, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, or psychotic disorder due to another medical condition
* Diagnosis of intellectual disability (IQ < 70).
* Participant has a history of meeting DSM-5 diagnosis for any substance-related disorder (except caffeine- and tobacco-related) within the 3 months before Visit 1.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in PANSS total score at Week 6 | Baseline to Week 6
  The Positive and Negative Syndrome Scale is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS total score is rated based on a structured clinical interview with the patient and supporting clinical information obtained from family, hospital staff, or other reliable informants. This assessment provides scores in 9 clinical domains, including a positive syndrome, a negative syndrome, depression, a composite index, and general psychopathology. Each item is scored on a 7-point (1 to 7) scale, with 1 being minimal impact, and 7 being highest impact. The cumulative score ranges from 30 to 210. A negative change from baseline score indicates improvement.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (9):
  - ProScience Research Group, Culver City, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Bloomfield Hills MI, Bloomfield Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - UB Department of Psychiatry, Buffalo, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
- Bulgaria (2):
  - Clinic of Child Psychiatry St. Nikolas, Sofia
  - MHAT Targovishte, Targovishte
- Colombia (5):
  - Centro de Investigaciones y Proyectos en Nerurociencia. CIPNA. IPS. SAS., Barranquilla
  - E.S.E. Hospital Mental de Antioquia, Bello
  - Centro de Investigacion del Sitema Nervioso CISNE, Bogotá
  - Instituto Colombiano Sistema Nervioso Clinica Monserrat, Bogotá
  - Psynapsis Salud Mental SA, Pereira
- Mexico (9):
  - Centro para la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Instituto de Investigacion Clinica AC, Durango
  - Consultorio de Medicina Especializada del Sector Privado, Guadalajara
  - Consultorio Medico En Psiquiatria de Niños y Adolescentes Hospital Aranda de la Parra, Guanajuato City
  - Medical Care and Research S.A. de C.V., Mérida
  - Iecsi S.C., Monterrey
  - CIT Neuropsique, Monterrey
  - Instituto de Informacion e Investigacion en Salud Mental AC, Monterrey
  - BLIND Investigaciones SC, San Luis Potosí City
- Romania (2):
  - Socola Psychiatric Institute Iasi, Iași
  - Spitalul Clinic de Urgenta Pentru Copii Louis Turcanu Clinica de Psihiatrie Copii Si Adolescenti, Timișoara
- Russia (19):
  - State Institution of Healthcare "Arkhangelsk Regional Clinical Psychiatric Hospital", Arkhangelsk
  - Kazan State Medical University KSMU, Kazan'
  - SBHI Specialized Clinical Psychiatric Hospital 1, Krasnodar
  - Regional Public Institution "Lipetsk Regional Psychoneurological Hospital", Lipetsk
  - Joint-Stock Company Scientific Centre of Personalized Medicine, Moscow
  - SBHI of Moscow Region "Central Clinical Psychiatric Hospital", Moscow
  - Clinical Psychiatry Hospital #1 of Nizhniy Novgorod, Nizhny Novgorod
  - State Public Institution of Healthcare Leningrad Regional Psychoneurological Dispensary, Roshchino
  - Saint-Petersburg GUZ Psychiatric Hospital No.1 n.a. P.P. Kaschenko, Saint Petersburg
  - Federal State Budgetary Institution "National Medical Research Center of Psychiatry and Neurology n.a. V.M. Bekhterev" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - Center for Medical Rehabilitation named after S.S. Mnukhin, Saint Petersburg
  - City Psychiatric Hospital #3 after I.I. Skvortsova-Stepanova, Saint Petersburg
  - GBUZ Samara Regional Clinical Psychiatric Hospital, Samara
  - State Budgetary Healthcare Institution "Saratov City Clinical Hospital #2 n.a. V.I. Razumovsky", Saratov
  - Smolensk State Medical University, Smolensk
  - LLC Podderzhka, Stavropol
  - LLC Clinic "Sto Let", Tomsk
  - Stavropol Regional Psychiatric hospital #2, Tonnel’nyy
  - Yaroslavl Regional Psychiatric Hospital, Yaroslavl Region
- Serbia (3):
  - Clinic.Neuro.Psych.Child.Youth, Belgrade
  - Institute for Mental Health, Belgrade
  - Clinic for psychiatry, KCV, Novi Sad
- Ukraine (8):
  - Regional Psychonevrological Hospital #3, Ivano-Frankivsk
  - SI "Institution of Neurology, Psychiatry and Narcology NAMS of Ukraine", Kharkiv
  - State Institution "Institute of Health Care for Children and Adolescents of the AMS of Ukraine, Kharkiv
  - Kherson Regional Institution of Mental Care, Kherson
  - SI Research Institute of Psychiatry of MoH of Ukraine, Kyiv
  - Communal Institution of Lviv Regional Council Lviv Regional Clinical Psychiatric Hospital, Lviv
  - Odesa Regional Medical Centre of Mental Health, Odesa
  - Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I. Yushchenko", Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Gedeon Richter will share de-identified patient-level data and study-level data for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. For more information please contact ra.ctarichter@richter.hu.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.